CLINICAL TRIAL: NCT01347034
Title: A Phase II Study Evaluating Neoadjuvant Administration of High Dose Radiation Therapy and Intratumoral Autologous Dendritic Cells in Patients With High-risk Soft Tissue Sarcomas
Brief Title: Radiation Therapy and Intratumoral Autologous Dendritic Cells in Soft Tissue Sarcomas (STS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16441
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: radiation; neoadjuvant; intratumoral; autologous; dendritic cells
MeSH Terms: conditions — Sarcoma | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Beam Radiation Therapy (RT) (Active Comparator): Arm A - University of Florida - External Beam Radiation Therapy (RT) - As outlined in Intervention Description
  Interventions: Procedure: External Beam Radiation Therapy (RT)
- External Beam RT + DC Injection (Experimental): Arm B - Moffitt Cancer Center - External Beam RT + Autologous Dendritic Cells (DC) Injection - As outlined in Intervention Description
  Interventions: Procedure: External Beam Radiation Therapy (RT); Biological: Autologous Dendritic Cells

INTERVENTIONS:
Procedure: External Beam Radiation Therapy (RT) — Day 1: Start external beam RT, 25 fractions from days 1-33 administered Monday through Friday only (no conventional external beam RT on days 6, 7, 13, 14, 20, 21, 27, or 28
  Days 57-70: Surgery will occur 3-5 weeks after the final dose of external beam RT.
  Day 78-91: First post-operative visit
  Days 91-365: Clinical follow-up
  Beyond day 365, follow-up will be conducted using the standard of care approach applicable to these patients for the determination of disease recurrence, progression and survival.
Biological: Autologous Dendritic Cells — Prior to each injection on Arm B, patients may receive prophylactic doses of a first generation cephalosporin antibiotic per physician discretion.
  Following each DC injection, Arm B patients will assess procedure-associated pain on a scale of 0-10. The next Monday following each DC injection, the patient will be called and questioned about such procedure associated toxicities.
  Other Names: immunotherapy
  Arms: External Beam RT + DC Injection

SUMMARY:
The purpose of this study is to determine if injection of the participant's our own immune related white blood cells (called dendritic cells) into their tumor will strengthen their immune system to fight against their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate or High grade (AJCC 7th edition Grade 3 and 4 or Grade 2 and 3 of a 3 tier system) STS as determined by local pathology diagnostic biopsy specimen review
* Musculoskeletal tumor in extremities, trunk or chest wall
* Primary tumor or isolated locally recurrent tumor greater than 5 cm in diameter as measured by Response Evaluation Criteria In Solid Tumors (RECIST) criteria v1.1
* Clinical Stage T2N0M0 (AJCC 7th edition)
* Age ≥18 years at time of consent
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0 or 1
* Patient's written study specific, Institutional Review Board (IRB) stamped informed consent.
* Adequate organ function (measured within a week prior to beginning treatment for Arm B and within 2 weeks of beginning treatment for Arm A): white blood count (WBC) > 3,000/mm³ and absolute neutrophil count (ANC) >1500/mm³; Platelets > 100,000/mm³; Hematocrit > 25%; Bilirubin < 2.0 mg/dL; Creatinine < 2.0 mg/dL, or creatinine clearance > 60 mL/min
* Radiation Oncologist must confirm that a 2-3 cm strip of skin can be spared from RT.

Exclusion Criteria:

* Retroperitoneal or Head and Neck primary locations
* Gastrointestinal stromal tumor (GIST)
* Demonstrated metastatic disease
* Contraindication to resection
* Prior RT if the current tumor is locally recurrent after prior resection
* Concurrent treatment with any anticancer agent other than RT as dictated by the protocol
* Prior chemotherapy for the pre-surgical treatment of the primary tumor (neoadjuvant chemotherapy)Bleeding/coagulation disorder
* Human Immunodeficiency Virus (HIV) infection or other primary immunodeficiency disorder
* Ongoing systemic therapy with immunosuppressant drugs (e.g. corticosteroids, azathioprine, cyclosporin, methotrexate)
* Steroid therapy within 4 weeks of first DC administration
* Any serious ongoing infection
* Pregnant or lactating women. Patients in reproductive age must agree to use contraceptive methods for the duration of the study (*A pregnancy test will be obtained before treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Daniel Indelicato, M.D., Principal Investigator — University of Florida, Shands Jacksonville
Locations (3):
- United States (3):
  - Shands University of Florida Department of Radiation Oncology, Gainesville, Florida
  - Shands Jacksonville Department of Radiation Oncology, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

REFERENCES:
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: External Beam Radiation Therapy (RT): Arm A - University of Florida - External Beam Radiation Therapy (RT) - As outlined in Intervention Description
- Experimental: External Beam RT + DC Injection: Arm B - Moffitt Cancer Center - External Beam RT + Autologous Dendritic Cells (DC) Injection - As outlined in Intervention Description
Period: Overall Study
Arm/Group | Active Comparator: External Beam Radiation Therapy (RT) | Experimental: External Beam RT + DC Injection
Started | 6 | 14
Completed | 6 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: External Beam Radiation Therapy (RT) | Experimental: External Beam RT + DC Injection | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Mean (Full Range); unit: years] | 53.8 [45 to 74] | 59.5 [42 to 77] | 57.35 [42 to 77]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 10 | 13
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 6 | 14 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Enhanced T Lymphocyte Immune Response Specific for Soft Tissue Sarcoma Tumor Associated Antigens(STS-TAAs)
Description: Investigate the ability of an intensified radiation therapy (RT) regimen (namely, conventional RT with a high-dose hypofractionated boost) and Dendritic Cell (DC) administration to induce an enhanced T lymphocyte immune response specific for STS-TAAs. Criteria for immune response evaluation: Individual patients were considered as responders to TAAs if at any time point the response in IFN-γ ELISPOT assay was found higher than 30 spots per 200,000 cells or in proliferation assay higher than 3000 counts/min (CPM) AND the response in IFN-γ ELISPOT or proliferation assays to tumor cell lysates (TCL) or Ad-Surv was found more than 2SD higher than the response to corresponding control lysate or Ad-c at the same time point AND 2SD higher than the response to the same stimuli at a base line (before start of the treatment).
Time Frame: 11 weeks per participant
Population: All participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: External Beam Radiation Therapy (RT) | Experimental: External Beam RT + DC Injection
Number analyzed (Participants) | 6 | 14
participants | 2 | 5

2. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: Evaluate the safety of intratumoral injections of DCs in combination with an intensified RT regimen patients with high-grade large STS. Toxicity assessments were performed weekly to include assessments for: constitutional symptoms, fever, fatigue; common radiation side effects; special attention was paid to DC injection and biopsy related toxicity. Only treatment related SAEs and AEs are reported for this measure.
Time Frame: 11 weeks per participant
Population: All participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: External Beam Radiation Therapy (RT) | Experimental: External Beam RT + DC Injection
Number analyzed (Participants) | 6 | 14
participants
  Treatment Emergent SAEs | 0 | 0
  Treatment Emergent Other AEs | 6 | 14

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Description: All adverse events, regardless of causality.
Arm/Group | Active Comparator: External Beam Radiation Therapy (RT) | Experimental: External Beam RT + DC Injection
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/14
Other Adverse Events (participants affected / at risk) | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: External Beam Radiation Therapy (RT) (N=6) | Experimental: External Beam RT + DC Injection (N=14)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Not related to therapy
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Not related to therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: External Beam Radiation Therapy (RT) (N=6) | Experimental: External Beam RT + DC Injection (N=14)
Fatigue (General disorders) | 2 (3) | 8 (11)
Pain (General disorders) | 3 (3) | 5 (11)
Edema limbs (General disorders) | 0 (0) | 4 (7)
Chills (General disorders) | 0 (0) | 1 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 11 (12)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 6 (11)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4)
Weight loss (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 7 (10)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Investigators planned to accrue 21 patients in each arm for a total of 42 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes